CLINICAL TRIAL: NCT05536427
Title: An Open-Label, Multi-Center, Multiple-Dose, Dose-Escalation and Dose-Expansion, Investigator-Initiated Phase I Clinical Study to Observe and Evaluate the Tolerability, Safety, Pharmacodynamics, and Preliminary Efficacy of IPM001 Injection in the Treatment of Progressive Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of IPM001 in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Immupeutics Medicine Technology Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-22PJ157
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPM001 (Experimental): A neoantigen/ tumor-specific antigen sencitized autoimmune cell injection
  Interventions: Biological: IPM001

INTERVENTIONS:
Biological: IPM001 — IPM001 will be used against tumor cells

SUMMARY:
In this study, safety and effects of IPM001 injection on human hepatocellular carcinoma are going to be investigated, IPM001 is a multiple tumor-associated antigen (TAA) and neoantigen/tumor-specific antigen (TSA) sensitized autoimmune cell injection

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and voluntarily sign the informed consent forms;
2. Subjects aged 18-75 years old (inclusive), male or female;
3. Subjects with progressive hepatocellular carcinoma who failed second-line therapy;
4. Subjects with an expected survival ≥ 6 months;
5. Subjects with a Child-Pugh score ≤ 7;
6. Subjects with an HLA A-02 genotype;
7. Subjects with a TBS score < 8;
8. Subjects with an ECOG score of 0-2 (inclusive);
9. Male and female subjects of childbearing potential must agree to use highly effective contraceptive methods during the entire study and for at least 3 months after receiving the last treatment, and women of childbearing age must have a negative pregnancy test;
10. Weight: Male > 50 kg, female > 45 kg;
11. Subjects with liver tumor lesions that can be used for tumor tissue biopsy. If feasible, the subjects must agree to provide tumor tissue specimens at baseline;
12. Subjects with no major organ dysfunctions (by laboratory test): ① white blood cell count ≥ 3.0 × 109/L; ② neutrophil count ≥ 1.5 × 109/L; ③ hemoglobin ≥ 90 g/L; ④ platelet count ≥ 30 × 109/L; ⑤ total bilirubin ≤ 2 × ULN; ⑥ Serum AST (GOT) and ALT (GPT) ≤ 2.5 × ULN; ⑦ albumin ≥ 3.0 g/dL (30 g/L); ⑧ blood creatinine ≤ 1.5 × ULN; ⑨ generally normal bleeding and coagulation time, with PT prolongation ≤ 4 s; ⑩ no serious cardiopulmonary diseases;
13. For subjects with hepatitis B-related primary hepatocellular carcinoma (HBV-HCC) or hepatitis C-related primary hepatocellular carcinoma (HCV-HCC), those who are with the following conditions are eligible to be enrolled:

    1. HBV-HCC: resolved HBV infection (specified as with positive HBV surface antibody and HBV core antibody, negative HBV surface antigen, and the HBV-DNA below the lower limit of detection); chronic HBV infection (specified as with positive HBV surface antigen or the HBV-DNA above the lower limit of detection, as well as the HBV-DNA less than 106 copies/mL), with concomitant antiviral therapy.
    2. HCV-HCC: resolved or active HCV infection (specified as with positive HCV antibody or the HCV-RNA above the lower limit of detection, as well as the HCV-RNA less than 103 copies/mL), where concomitant antiviral therapy may be given for active HCV infection.
14. Subjects with no obvious genetic diseases;
15. Subjects who have not received any live attenuated vaccines within 4 weeks prior to the first administration;
16. Subjects who are able to follow the clinical study protocol and follow-up procedures.

Exclusion Criteria:

1. Subjects with immunodeficiency or a history of autoimmune disorders (e.g., rheumatoid arthropathy, systemic lupus erythematosus, vasculitis, multiple sclerosis, insulin-dependent diabetes mellitus, etc.);
2. Subjects with severe concurrent medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes mellitus, uncontrolled hypertension, serious infection and infectious disease, active peptic ulcer, presence of active hemorrhage, and severe organ failure;
3. Subjects with myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, Grade III or IV cardiac failure defined by the New York Heart Association (NYHA), epileptic seizure, and mechanical or paralytic ileus within 6 months prior to the first administration of the investigational drug;
4. Subjects who have received chemotherapy and hormonal therapy within 28 days prior to signing the informed consent forms, or are currently taking other investigational drugs;
5. Subjects with lymphoma, leukemia, myelodysplastic syndrome (MDS), or myelosuppression;
6. Subjects with allergy or a history of hypersensitivity to human blood albumin, or a history of allergy or hypersensitivity to any investigational drug or its excipients;
7. Subjects with chronic diseases requiring immunotherapy or hormonal therapy; and subjects currently receiving corticosteroids for other diseases (except those using topical or inhaled steroids);
8. Pregnant or lactating women;
9. Subjects with mental or neurological disorders that are not easily controlled;
10. Subjects infected with human immunodeficiency virus (commonly known as AIDS) or treponema pallidum (commonly known as syphilis);
11. Subjects with a history of other malignant tumors within the last 5 years;
12. Subjects with prior allogeneic stem cell transplantation or solid organ transplant;
13. Subjects with a history of drug or alcohol abuse;
14. Subjects with any irAE of ≥ Grade 3 following prior immunotherapy;
15. Subjects who, in the judgment of the investigator, are not suitable to participate in this clinical study (e.g., with poor compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
safety (AE/ irAE/ SAE) | 12 months
  Adverse events, Immue-related adverse，serious adverse event
Tolerance(DLT/ MTD/ OBD) | 12 months
  Dose Limiting Toxicity, Maximum Tolerated Dose, Optimal Biological Dose

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 12 months
  The time between the NeoAg/aeTSA CTL initiation and the onset of tumor progress or death from any cause
Overall Survival (OS) | 12 months
  From the beginning of NeoAg/aeTSA CTL initiation to the time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No